CLINICAL TRIAL: NCT00665652
Title: A Phase II Trial of Lenalidomide as a Treatment for Neuropathy Associated With Nonmalignant Monoclonal Gammopathy of Undetermined Significance (MGUS)
Brief Title: Study of Lenalidomide as a Treatment for Neuropathy Associated With Monoclonal Gammopathy of Undetermined Significance
Acronym: MGUS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study has been suspended for slower than anticipated enrollment to date.
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Principal Investigator, Elijah W. Stommel, MD, PhD, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RV-PN-PI-235 D0713
Record Dates: First submitted 2008-04-22; First posted 2008-04-24 (Estimated); Results first posted 2018-09-11 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-08

CONDITIONS: Neuropathy; Nonmalignant Monoclonal Gammopathy of Undetermined Significance (MGUS)
Keywords: Neuropathy; Nonmalignant Monoclonal Gammopathy of Undetermined Significance (MGUS); MGUS
MeSH Terms: interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide (Experimental)
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — Subjects will receive lenalidomide 25 mg per day for days 1-21 followed by 7 days rest (28-day cycle) for 12 cycles.

SUMMARY:
The purpose of the study is to learn about the effects of the drug, lenalidomide (Revlimid®), on neuropathy (damage to the nerves that affect feelings and strength) associated with Nonmalignant Monoclonal Gammopathy of Undetermined Significance (MGUS).

DETAILED DESCRIPTION:
Screening:

All subjects eligible for screening must sign an informed consent for the study prior to any study related procedures.

Study Design:

This is an open-label, single-institutional clinical study of lenalidomide as a treatment for MGUS associated neuropathy. Eligible patients will be followed for 28 days before starting study drug. Subjects who remain eligible during the 28 day pretreatment period will receive lenalidomide 25 mg per day for days 1-21 followed by 7 days rest (28-day cycle) for 12 cycles. All patients on treatment will be followed and will be included in the intention to treat group. Patients will be evaluated every three months with the TNS. On-treatment patients must come to clinic at least monthly for the first 3 cycles, and then can come as per the schedule of study assessments only if they are on a stable dose of lenalidomide for at least one cycle. Subjects will be enrolled in the study for up to 14 months.

Lenalidomide administration:

Lenalidomide is an oral medication that will be taken at approximately the same time each day with or without food.

Lenalidomide capsules should be swallowed whole, and should not be broken, chewed or opened.

If a dose of lenalidomide is missed, it should be taken as soon as possible on the same day. If it is missed for the entire day, it should not be made up.

Patients who take more than the prescribed dose of lenalidomide should be instructed to seek emergency medical care if needed and contact study staff immediately.

Dosing Regimen:

The planned dose of lenalidomide for investigation is 25 mg/day, orally on days 1-21 followed by 7 days rest (28 day cycle). Dosing will be in the morning at approximately the same time each day. The planned dose is: Plavix 75mg/day or aspirin 325mg/day.

Subjects experiencing adverse events may need study treatment modifications

ELIGIBILITY:
Inclusion Criteria:

* Clinically proven MGUS associated neuropathy with a Total Neuropathy Score (TNS) ≥5 (determined by exam, history and confirmatory EDX testing in association with MGUS (IgM,IgG,IgA))
* Disease duration less than or equal to 8 years
* Able to take Plavix 75mg/day or aspirin 325 mg daily as prophylactic anticoagulation. (patients currently taking warfarin with a stable INR may stay on current dose)

Exclusion Criteria:

* Patients previously treated with thalidomide
* Patients previously treated with lenalidomide
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs
* Known positive for HIV or infectious hepatitis, type A, B or C
* Medical history of deep venous thrombosis or hyper-coagulable state
* Gastrointestinal abnormalities including: inability to take oral medication, requirement for intravenous alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease
* Patients with dementia, other serious neurological diseases, uncompensated medical illness, substance abuse and debilitating psychiatric illness.
* A serious uncontrolled medical disorder or active infection that would impair the patient's ability to receive study treatment. Significant cardiac disease, including uncontrolled high blood pressure, unstable angina, congestive heart failure, myocardial infarction within the previous 6 months or serious cardiac arrhythmias will be excluded.
* Medical conditions associated with neuropathy such as active thyroid disease, diabetes mellitus, and lupus, nutritional deficiencies, malignancy, human immunodeficiency virus infection, alcohol dependence, amyloidosis, or connective tissue diseases and Guillain-Barre Syndrome. Medications or toxic exposures known to cause neuropathy, or a family history of neuropathy will also be grounds for exclusion.
* Pregnant or breast feeding females. (Lactating females must agree not to breast feed while taking lenalidomide).
* Subjects who are allergic to aspirin or Plavix (clopidogrel)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2008-04; Primary Completion 2011-05-19 (Actual); Study Completion 2011-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elijah W. Stommel, MD, PhD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lenalidomide
Started | 8
Completed | 2
Not Completed | 6
Not completed — Adverse Event | 4
Not completed — Death | 1
Not completed — No longer met inclusion criteria. | 1

BASELINE CHARACTERISTICS:
Arm/Group | Lenalidomide
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Neuropathy Score in Subjects With MGUS Associated Neuropathy After Treatment With Lenalidomide.
Description: Minimum value of the Total Neuropathy Score is "0", maximum value is "40". A higher score represents a worsening.
Time Frame: Baseline, 12 months
Population: Subjects were evaluable if they were on study drug for 3 months.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Lenalidomide
Number analyzed (Participants) | 6
units on a scale | 0.17 [-4 to 5]

ADVERSE EVENTS:
Time Frame: Informed consent obtained through Month 14.
Arm/Group | Lenalidomide
All-Cause Mortality (participants affected / at risk) | 1/8
Serious Adverse Events (participants affected / at risk) | 3/8
Other Adverse Events (participants affected / at risk) | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide (N=8)
Ischemic Colitis (Gastrointestinal disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes